CLINICAL TRIAL: NCT01768910
Title: The Bladder and the Brain - Investigation of the Supraspinal Neural Control of Lower Urinary Tract Function in Healthy Subjects and Patients With Neurogenic and Non-neurogenic Bladder Dysfunction Using Advanced Neuroimaging Techniques
Brief Title: Supraspinal Control of Lower Urinary Tract Function in Healthy Controls and Patients With Bladder Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH-2011-0346/PB_2016-00872
Record Dates: First submitted 2013-01-08; First posted 2013-01-16 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Neurogenic Lower Urinary Tract Dysfunction; Multiple Sclerosis; Overactive Bladder; Spinal Cord Injury
Keywords: lower urinary tract; bladder; supraspinal control; neuroimaging; functional magnetic resonance imaging; diffusion tensor imaging; functional connectivity; neurogenic lower urinary tract dysfunction; overactive bladder; multiple sclerosis; spinal cord injury
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy controls (Experimental): Procedure: 1-2 fMRI measurements within 4 weeks from first exam. Measurements include repetitive retrograde bladder filling via transurethral catheter at different bladder volumes and temperatures (e.g. bladder cooling, body warm or room temperature)of the filling liquid.
  Interventions: Other: fMRI; Other: bladder filling; Other: bladder cooling
- MS with OAB (Experimental): Procedure: 1-2 fMRI measurements within 4 weeks from first exam. Measurements include repetitive retrograde bladder filling via transurethral catheter at different bladder volumes and temperatures of the filling liquid.
  Interventions: Other: fMRI; Other: bladder filling; Other: bladder cooling
- MS without OAB (Experimental): Procedure: 1-2 measurements within 4 weeks from first exam. Measurements include repetitive bladder filling via transurethral catheter at different bladder volumes and temperatures of the filling liquid.
  Interventions: Other: fMRI; Other: bladder filling; Other: bladder cooling
- NNOAB (Experimental): Procedure: 1-2 measurements within 4 weeks from first exam. Measurements include repetitive bladder filling via transurethral catheter at different bladder volumes and temperatures of the filling liquid plus additional post-treatment fMRI scan 5 to 7 weeks after OAB treatment (such as antimuscarinics, intradetrusor injections of botulinum toxin type A)
  Interventions: Other: fMRI; Other: bladder filling; Other: bladder cooling; Other: additional post-treatment fMRI scan
- SCI with neurogenic detrusor overactivity (Experimental): Procedure: 1-2 measurements within 4 weeks from first exam. Measurements include repetitive bladder filling via transurethral catheter at different bladder volumes and temperatures of the filling liquid plus 1 additional post-treatment fMRI scan 5 to 7 weeks after intradetrusor injections of botulinum toxin type A
  Interventions: Other: fMRI; Other: bladder filling; Other: bladder cooling; Other: additional post-treatment fMRI scan

INTERVENTIONS:
Other: fMRI — 2 measurements using functional magnetic resonance imaging in a 3T scanner
Other: bladder filling — Repetitive retrograde bladder filling via transurethral catheter with different filling volumes using body warm saline during each of the fMRI measurements.
Other: bladder cooling — Retrograde bladder filling via transurethral catheter with 4-8°C saline during each of the fMRI measurements.
Other: additional post-treatment fMRI scan — Should NNOAB or SCI patients receive a study independent OAB therapy by their treating physician after the 2nd fMRI scan, they will be invited for an additional third fMRI scan.
  Arms: NNOAB; SCI with neurogenic detrusor overactivity

SUMMARY:
The purpose of this study is to provide profound insight into the supraspinal neuronal mechanisms and networks responsible for lower urinary tract (LUT) control and to verify, amend or adjust neuronal circuitry models established from findings in healthy subjects in the context of neurogenic and non-neurogenic LUT dysfunction.

DETAILED DESCRIPTION:
The subject recruitment will be performed within the Neuro-Urology outpatient clinic at the Balgrist University Hospital and in collaboration with the Departments of Neurology, Urology and Gynecology at the University Hospital Zürich.

The following subject groups will be recruited: 1) healthy controls (n=22), Non-neurogenic overactive bladder (NNOAB) patients (n=20), multiple sclerosis (MS) patients with OAB (n=15), MS patients without OAB (n=15), spinal cord injury (SCI) patients with neurogenic detrusor overactivity (n=24).

After inclusion, all subjects and patients will undergo one to two functional magnetic resonance imaging (fMRI) sessions. NNOAB patients might undergo an additional fMRI session after receiving overactive bladder (OAB) treatment (such as antimuscarinics, intradetrusor injections of botulinum toxin type A). Spinal cord injury (SCI) patients with neurogenic detrusor overactivity will undergo an additional fMRI session 5-7 weeks after intradetrusor injections of botulinum toxin type A.

High-resolution anatomical images and functional blood-oxygen-level-dependent (BOLD)-signal sensitive images will be acquired. In addition to the fMRI, diffusion tensor imaging (DTI) sequences will be recorded after the anatomical scans to provide information about the structural supraspinal connectivity.

Study endpoints are changes of the BOLD signal in regard to location and intensity, structural and functional connectivity (FC) between previously described supraspinal centers involved in LUT control, and statistical differences of changes in BOLD signals, structural and functional connectivity between patients and healthy controls.

All acquired fMRI data will be transferred to an off-line workstation running BrainVoyager QX or Statistical Parametric Mapping (SPM) Version 8. The functional data will be pre-processed for motion correction, spatial smoothing, linear trend removal, and temporal high-pass filtering. With both programs statistical analysis and graphical presentation of the results can be performed.

The DTI records will be evaluated with SPM8, BrainVoyager QX or other programs like Functional Magnetic Resonance Imaging of the Brain (FMRIB) Software Library (FSL) and DTI-Studio. To estimate FC we will use SPM8 or the brain connectivity toolbox. Both softwares allow the estimation of rest- and task-related connectivity on single subject and group level with corrected statistical threshold.

Overall, 96 subjects for the main study are estimated to be sufficient to demonstrate significant differences between groups.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

* Right handed
* MR suitability
* Written informed consent
* unimpaired LUT function

MS patients with OAB

* Right handed
* MR suitability
* Written informed consent
* diagnosis of MS according to the McDonald criteria
* Expanded Disability Status Scale (EDSS) ≤ 6
* OAB symptoms since > 6 months

  * ≥ 3 episodes of urinary urgency
  * frequency > 8/24h
* with or without detrusor overactivity

MS patients without OAB

* Right handed
* MR suitability
* Written informed consent
* diagnosis of MS according to the McDonald criteria
* Expanded Disability Status Scale (EDSS) ≤ 6

Patients with NNOAB

* Right handed
* MR suitability
* Written informed consent
* idiopathic OAB symptoms since > 6 months

  * ≥ 3 episodes of urinary urgency
  * frequency > 8/24h
* refractory to antimuscarinic treatment for ≥ 1 month
* indication for intradetrusor injections of Botulinumtoxin Type A
* willingness and ability to perform self-catheterization

SCI patients with neurogenic detrusor overactivity

* Right handed
* MR suitability
* Written informed consent
* neurogenic detrusor overactivity due to SCI
* indication for intradetrusor injections of botulinum toxin type A

Exclusion Criteria:

Healthy controls

* impaired LUT function
* pregnancy or breast feeding
* no informed consent
* any craniocerebral injury or surgery
* any permanent ferromagnetic implant
* any previous surgery of the LUT or genitalia
* any anatomical anomaly of the LUT or genitalia
* any LUT malignancy
* postvoid residual urine volume (PVR) > 150ml
* current urinary tract infection
* any LUT symptoms

  * ≥ 3 episodes of urinary urgency
  * frequency > 8/24h

MS patients with OAB

* pregnancy or breast feeding
* any permanent ferromagnetic implant
* any neurological or psychological disease despite MS
* any craniocerebral injury or surgery
* any previous surgery of the LUT or genitalia
* any anatomical anomaly or malignancy of the LUT or genitalia
* any metabolic disease
* PVR > 150ml
* any concomitant treatment for the LUT (e.g. neuromodulation)
* Stress urinary incontinence
* any condition other than MS that might explain OAB symptoms
* current urinary tract infection
* indwelling catheters or the necessity to perform self-catheterization

MS patients without OAB

* pregnancy or breast feeding
* any permanent ferromagnetic implant
* any neurological or psychological disease despite MS
* any craniocerebral injury or surgery
* any previous surgery of the LUT or genitalia
* any anatomical anomaly or malignancy of the LUT or genitalia
* any metabolic disease
* PVR > 150ml
* any concomitant treatment for the LUT (e.g. neuromodulation)
* Stress urinary incontinence
* any LUT symptoms

  * ≥ 3 episodes of urinary urgency
  * frequency > 8/24h
* indwelling catheters or the necessity to perform self-catheterization
* detrusor overactivity
* current urinary tract infection

Patients with NNOAB

* pregnancy or planned within next 8 months, breast feeding
* any permanent ferromagnetic implant
* any neurological, psychological, metabolic or cardiovascular disease
* any craniocerebral injury or surgery
* any previous surgery of the LUT or genitalia within the last year or that is related to the OAB symptoms
* any anatomical anomaly or malignancy of the LUT or genitalia
* PVR > 150ml
* Stress urinary incontinence
* indwelling catheters or the necessity to perform self-catheterization
* any concomitant treatment for the LUT (e.g. neuromodulation)
* current urinary tract infection

SCI patients with neurogenic detrusor overactivity

* pregnancy or breast feeding
* any permanent ferromagnetic implant
* any neurological or psychological disease despite SCI
* any craniocerebral injury or surgery
* any previous surgery of LUT of genitalia
* any anatomical anomaly or malignancy of the LUT or genitalia
* any metabolic disease
* any concomitant treatment for the LUT (e.g. neuromodulation)
* current urinary tract infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-07-17 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Bold signal | baseline and 4 weeks
  During fMRI measurements the changes of BOLD signal intensity in respect to certain supraspinal areas (e.g. pons, insula, anterior cingulate cortex, thalamus, supplementary motor area, prefrontal cortex) will be evaluated.
  Variables are age, bladder volume, urgency and attention.
Structural and functional connectivity | baseline and after potential OAB treatment
  Acquired data from the above mentioned measurements will be used to analyze structural and functional connectivity between supraspinal areas involved in the LUT control, especially between prefrontal, thalamus, insula, and anterior cingulate cortex.
  Variables are age, bladder volume, urgency and attention. Correlations of neuronal activity from the fMRI-data will be estimated using SPM8, brain connectivity tool box.

SECONDARY OUTCOMES:
Side effects | 3 years
  Pain, Lower urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mehnert, MD, Principal Investigator — Neuro-Urology, Spinal Cord Injury Center & Research, University of Zurich, Balgrist University Hospital, Forchstrasse 340, 8008 Zurich, Switzerland; Thomas M Kessler, MD, Principal Investigator — Neuro-Urology, Spinal Cord Injury Center & Research, University of Zurich, Balgrist University Hospital, Forchstrasse 340, 8008 Zurich, Switzerland; Spyros Kollias, MD, Principal Investigator — Institute of Neuroradiology, University Hospital Zurich, Sternwartstrasse 6, 8091 Zurich, Switzerland
Locations (2):
- Switzerland (2):
  - Neuro-Urology, Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital, Zurich
  - University Hospital Zürich, Zurich

REFERENCES:
- [Result] Walter M, Michels L, Kollias S, van Kerrebroeck PE, Kessler TM, Mehnert U. Protocol for a prospective neuroimaging study investigating the supraspinal control of lower urinary tract function in healthy controls and patients with non-neurogenic lower urinary tract symptoms. BMJ Open. 2014 May 21;4(5):e004357. doi: 10.1136/bmjopen-2013-004357. PMID 24848086
- [Result] Leitner L, Walter M, Freund P, Mehnert U, Michels L, Kollias S, Kessler TM. Protocol for a prospective magnetic resonance imaging study on supraspinal lower urinary tract control in healthy subjects and spinal cord injury patients undergoing intradetrusor onabotulinumtoxinA injections for treating neurogenic detrusor overactivity. BMC Urol. 2014 Aug 18;14:68. doi: 10.1186/1471-2490-14-68. PMID 25132340
- [Result] Leitner L, Walter M, Jarrahi B, Wanek J, Diefenbacher J, Michels L, Liechti MD, Kollias SS, Kessler TM, Mehnert U. A novel infusion-drainage device to assess lower urinary tract function in neuro-imaging. BJU Int. 2017 Feb;119(2):305-316. doi: 10.1111/bju.13655. Epub 2016 Oct 20. PMID 27617867
- [Result] Walter M, Leitner L, Michels L, Liechti MD, Freund P, Kessler TM, Kollias S, Mehnert U. Reliability of supraspinal correlates to lower urinary tract stimulation in healthy participants - A fMRI study. Neuroimage. 2019 May 1;191:481-492. doi: 10.1016/j.neuroimage.2019.02.031. Epub 2019 Feb 15. PMID 30776530